CLINICAL TRIAL: NCT01362946
Title: Designing a Novel Behavioral Treatment Protocol for Children Characterized by Conduct Problems and Callous-unemotional Traits
Brief Title: Behavioral Treatment for Children With Conduct Problems and Callous-Unemotional Traits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1R34MH085796-01A2 (NIH); 1R34MH085796-01A2 (NIH)
Record Dates: First submitted 2011-01-07; First posted 2011-06-01 (Estimated); Results first posted 2016-01-15 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2015-12

CONDITIONS: Conduct Disorder; Oppositional Defiant Disorder
Keywords: Conduct problems; callous-unemotional traits; disruptive behavior disorders
MeSH Terms: conditions — Conduct Disorder; Oppositional Defiant Disorder; Attention Deficit and Disruptive Behavior Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reward-Emphasized treatment (Experimental): This treatment consisted of behavior therapy modified to match the unique learning styles of children with CPCU. This was accomplished by emphasizing rewards and de-emphasizing punishments. This treatment was administered using a summer treatment program.
  Interventions: Behavioral: Reward-Emphasized Treatment
- Standard treatment (Active Comparator): This treatment consisted of standard behavior therapy, in which reward and punishment components were used in a balanced manner, as is typically done in outpatient settings. This treatment was administered using a summer treatment program.
  Interventions: Behavioral: Standard Treatment

INTERVENTIONS:
Behavioral: Reward-Emphasized Treatment — Intensive behavioral treatment delivered in a summer camp setting, with reward components emphasized and punishment components de-emphasized
  Arms: Reward-Emphasized treatment
Behavioral: Standard Treatment — Intensive behavioral treatment delivered in a summer camp setting, with rewards and punishment equally emphasized.
  Arms: Standard treatment

SUMMARY:
The purpose of this study is to modify behavior therapy so that it is optimized for children with conduct problems and callous-unemotional traits by emphasizing reward components and de-emphasizing punishment components.

DETAILED DESCRIPTION:
Several studies have demonstrated that standard behavioral treatments do not appear to be sufficient for children with conduct problems (CP) and callous-unemotional (CU) traits. Other research suggests that children with CPCU are less responsive to punishments as evaluated using controlled laboratory tasks. Based on these two sets of findings, it was hypothesized that behavioral treatment modified to emphasize reward and de-emphasize punishments would be advantageous when used to treat children with CPCU. This hypothesis was tested in a treatment development study that had three phases. During phase 1, which occurred in 2010, the intervention was planned and treatment procedures and manuals were developed. During phase 2, which occurred in 2011, a pilot study was conducted in which the intervention was tested in an iterative manner in a group of 12 children with conduct problems and callous-unemotional traits. In phase 3, a larger trial was conducted using a cross over design, with one-half of participants getting standard behavioral treatment for four weeks followed by modified behavioral treatment for four weeks and remaining participants receiving treatments in the reverse order.Treatments were evaluated using parent ratings, counselor ratings, and frequency counts of behavior during treatments.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of oppositional defiant disorder or conduct disorder
* Ages 7 to 12 years old
* t-score of 65 or above on CU scale of Antisocial Process Screening Device as rated by parents or teacher
* at least parent/caregiver fluent in English
* able to participate in vigorous outdoor activities
* parent/caregiver agreement to keep psychoactive medication treatment constant throughout the study

Exclusion Criteria:

* Full scale intelligence quotient (IQ) of less than 75
* medical conditions that contra-indicate participation in treatment
* current or past clinical diagnosis of pervasive developmental disorder, schizophrenia or other psychotic disorders, sexual disorder, organic mental disorder, or eating disorder
* lack of functional impairment
* current or past seizures or other neurological disorders

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Waschbusch, Ph.D., Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Modified Behavior Treatment Then Standard Behavior Treatment: Summer treatment program: Intensive behavioral treatment delivered in a summer camp setting. During the first four weeks, participants received modified behavioral treatment (MBT) that emphasized rewards and de-emphasized punishments. During the last four weeks, participants received standard behavior treatment (SBT) that balanced reward and punishment.
- Standard Behavior Treatment Then Modified Behavior Treatment: Summer treatment program: Intensive behavioral treatment delivered in a summer camp setting. During the first four weeks, participants received standard behavior treatment (SBT) that balanced reward and punishment. During the last four weeks of treatment, participants received modified behavioral treatment (MBT) that emphasized rewards and de-emphasized punishments.
Period: First Behavior Modification Block
Arm/Group | Modified Behavior Treatment Then Standard Behavior Treatment | Standard Behavior Treatment Then Modified Behavior Treatment
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0
Period: Second Behavior Modification Block
Arm/Group | Modified Behavior Treatment Then Standard Behavior Treatment | Standard Behavior Treatment Then Modified Behavior Treatment
Started | 23 (1 participant withdrew after last but before this treatment period - illness unrelated to study.) | 24
Completed | 23 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Sample: Summer treatment program: Intensive behavioral treatment delivered in a summer camp setting. During one block of four weeks, participants received modified behavioral treatment (MBT) that emphasized rewards and de-emphasized punishments. During another block of four weeks, participants received standard behavior treatment (SBT) that balanced reward and punishment. Order of treatment blocks was counter-balanced across participants, and primary analyses were within-subject comparisons. Therefore, we report demographics for the full sample.
Arm/Group | Overall Sample
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 48
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.29 (1.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 34
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Conduct Problems
Description: Counselors recorded each instance of conduct problems, defined as lying, stealing, intentional destruction of property, and intentional aggression. The average number per day was computed for each week of treatment.
Time Frame: Weekly
Population: Three children excluded from analyses; two excluded because of medication changes during treatment. One excluded because he was mistakenly enrolled (after collecting treatment data we learned that he did not meet all inclusion criteria).
Measure: Least Squares Mean (Standard Error); unit: Number of conduct problems per day
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
Number of conduct problems per day
  Standard Behavior Therapy - week 1 | 0.76 (0.27)
  Standard Behavior Therapy - week 2 | 1.08 (0.35)
  Standard Behavior Therapy - week 3 | 0.41 (0.54)
  Standard Behavior Therapy - week 4 | 0.92 (0.48)
  Modified Behavior Therapy - week 1 | 0.76 (0.28)
  Modified Behavior Therapy - week 2 | 1.26 (0.36)
  Modified Behavior Therapy - week 3 | 1.54 (0.54)
  Modified Behavior Therapy - week 4 | 1.42 (0.49)

2. Secondary Outcome: IOWA Inattentive/Overactive Scale - Counselor
Description: At the end of each treatment week counselors rated each child's overall inattentive-overactive-impulsive behavior during the week. Rating were completed using Likert scales that ranged from 0 ("not at all") to 3 ("very much"). Items were summed to compute a scale score with a theoretical range of 0 to 15.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
units on a scale
  Standard Behavior Therapy - week 1 | 5.36 (0.57)
  Standard Behavior Therapy - week 2 | 5.57 (0.58)
  Standard Behavior Therapy - week 3 | 6.15 (0.60)
  Standard Behavior Therapy - week 4 | 5.78 (0.58)
  Modified Behavior Therapy - week 1 | 5.51 (0.58)
  Modified Behavior Therapy - week 2 | 5.59 (0.58)
  Modified Behavior Therapy - week 3 | 5.95 (0.60)
  Modified Behavior Therapy - week 4 | 6.14 (0.58)

3. Primary Outcome: Negative Verbalizations
Description: Counselors recorded each instance of negative verbalizations, defined as verbal abuse to staff, teasing peers, and swearing. The average number per day was computed for each week of treatment.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number of negative verbals per day
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
Number of negative verbals per day
  Standard behavior therapy - week 1 | 5.70 (1.31)
  Standard behavior therapy - week 2 | 7.32 (1.53)
  Standard behavior therapy - week 3 | 6.73 (2.41)
  Standard behavior therapy - week 4 | 5.91 (1.98)
  Modified Behavior Therapy - week 1 | 4.94 (1.36)
  Modified Behavior Therapy - week 2 | 9.16 (1.58)
  Modified Behavior Therapy - week 3 | 10.63 (2.45)
  Modified Behavior Therapy - week 4 | 10.95 (2.01)

4. Primary Outcome: Complaining
Description: Counselors recorded each instance of complaining. The average number per day was computed for each week of treatment.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number of complaints per day
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
Number of complaints per day
  Standard Behavior Therapy - week 1 | 5.25 (1.02)
  Standard Behavior Therapy - week 2 | 4.92 (1.25)
  Standard Behavior Therapy - week 3 | 2.76 (1.32)
  Standard Behavior Therapy - week 4 | 3.54 (1.21)
  Modified behavior therapy - week 1 | 3.33 (1.00)
  Modified behavior therapy - week 2 | 5.18 (1.25)
  Modified behavior therapy - week 3 | 5.90 (1.32)
  Modified behavior therapy - week 4 | 5.95 (1.24)

5. Primary Outcome: Interruption
Description: Counselors recorded each instance of interrupting. The average number per day was computed for each week of treatment.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number of interruptions per day
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
Number of interruptions per day
  Standard Behavior Therapy - week 1 | 9.86 (1.32)
  Standard Behavior Therapy - week 2 | 14.81 (2.02)
  Standard Behavior Therapy - week 3 | 13.43 (2.51)
  Standard Behavior Therapy - week 4 | 12.61 (2.27)
  Modified Behavior Therapy - week 1 | 10.21 (1.41)
  Modified Behavior Therapy - week 2 | 14.32 (2.06)
  Modified Behavior Therapy - week 3 | 19.32 (2.54)
  Modified Behavior Therapy - week 4 | 19.66 (2.28)

6. Primary Outcome: Noncompliance
Description: Counselors recorded each instance of noncompliance. The average number per day was computed for each week of treatment.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number of noncompliance per day
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
Number of noncompliance per day
  Standard Behavior Therapy - week 1 | 3.82 (0.89)
  Standard Behavior Therapy - week 2 | 4.29 (0.97)
  Standard Behavior Therapy - week 3 | 3.52 (0.84)
  Standard Behavior Therapy - week 4 | 2.99 (0.85)
  Modified Behavior Therapy - week 1 | 3.35 (0.90)
  Modified Behavior Therapy - week 2 | 5.16 (0.97)
  Modified Behavior Therapy - week 3 | 4.26 (0.87)
  Modified Behavior Therapy - week 4 | 4.28 (0.87)

7. Primary Outcome: Rule Violations
Description: Counselors recorded each instance of rule violations. The average number per day was computed for each week of treatment.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number of rule violations per day
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
Number of rule violations per day
  Standard Behavior Therapy - week 1 | 36.65 (6.08)
  Standard Behavior Therapy - week 2 | 40.84 (6.10)
  Standard Behavior Therapy - week 3 | 33.93 (6.80)
  Standard Behavior Therapy - week 4 | 35.31 (7.26)
  Modified Behavior Therapy - week 1 | 27.28 (6.13)
  Modified Behavior Therapy - week 2 | 41.89 (6.06)
  Modified Behavior Therapy - week 3 | 46.99 (6.86)
  Modified Behavior Therapy - week 4 | 49.56 (7.21)

8. Primary Outcome: Positive Peer Behavior
Description: Counselors recorded each instance of positive behavior with peers, defined as helping, sharing and ignoring teasing. The average number per day was computed for each week of treatment.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number of positive peer behave per day
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
Number of positive peer behave per day
  Standard Behavior Therapy - week 1 | 4.91 (0.48)
  Standard Behavior Therapy - week 2 | 4.51 (0.48)
  Standard Behavior Therapy - week 3 | 4.84 (0.58)
  Standard Behavior Therapy - week 4 | 4.33 (0.49)
  Modified Behavior Therapy - week 1 | 5.42 (0.49)
  Modified Behavior Therapy - week 2 | 7.08 (0.51)
  Modified Behavior Therapy - week 3 | 6.72 (0.59)
  Modified Behavior Therapy - week 4 | 9.72 (0.52)

9. Primary Outcome: Minutes in Time Out
Description: Counselors recorded the total number of minutes children were in Time Out due to intentional aggression, intentional destruction of property, or repeated noncompliance. The average number per day was computed for each week of treatment.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Minutes in Time Out per day
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
Minutes in Time Out per day
  Standard Behavior Therapy - week 1 | 10.62 (3.03)
  Standard Behavior Therapy - week 2 | 14.77 (3.68)
  Standard Behavior Therapy - week 3 | 9.50 (3.33)
  Standard Behavior Therapy - week 4 | 10.17 (3.45)
  Modified Behavior Therapy - week 1 | 6.57 (3.06)
  Modified Behavior Therapy - week 2 | 12.15 (3.72)
  Modified Behavior Therapy - week 3 | 10.76 (3.45)
  Modified Behavior Therapy - week 4 | 10.67 (3.52)

10. Primary Outcome: Number of Time Outs
Description: Counselors recorded the total number of Time Outs children served due to intentional aggression, intentional destruction of property, or repeated noncompliance. The average number per day was computed for each week of treatment.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number of Time Outs per day
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
Number of Time Outs per day
  Standard Behavior Therapy - week 1 | 0.69 (0.25)
  Standard Behavior Therapy - week 2 | 1.00 (0.26)
  Standard Behavior Therapy - week 3 | 1.15 (0.28)
  Standard Behavior Therapy - week 4 | 0.76 (0.27)
  Modified Behavior Therapy - week 1 | 0.82 (0.27)
  Modified Behavior Therapy - week 2 | 1.09 (0.26)
  Modified Behavior Therapy - week 3 | 0.98 (0.28)
  Modified Behavior Therapy - week 4 | 1.27 (0.28)

11. Primary Outcome: Minutes of Physical Management
Description: Counselors recorded the total number of minutes children had to be physically managed due to behavior dangerous to themselves or others. The average number per day was computed for each week of treatment.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Minutes of Physical Manage per day
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
Minutes of Physical Manage per day
  Standard Behavior Therapy - week 1 | 0.09 (0.30)
  Standard Behavior Therapy - week 2 | 0.21 (0.16)
  Standard Behavior Therapy - week 3 | 0.29 (0.17)
  Standard Behavior Therapy - week 4 | 0.31 (0.17)
  Modified Behavior Therapy - week 1 | 0.54 (0.30)
  Modified Behavior Therapy - week 2 | 0.30 (0.16)
  Modified Behavior Therapy - week 3 | 0.28 (0.17)
  Modified Behavior Therapy - week 4 | 0.21 (0.17)

12. Secondary Outcome: IOWA Inattentive/Overactive Scale - Parent
Description: At the end of each treatment week parents rated each child's overall inattentive-overactive-impulsive behavior during the week. Rating were completed using Likert scales that ranged from 0 ("not at all") to 3 ("very much"). Items were summed to compute a scale score with a theoretical range of 0 to 15.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
units on a scale
  Standard Behavior Therapy - week 1 | 6.71 (0.59)
  Standard Behavior Therapy - week 2 | 7.11 (0.60)
  Standard Behavior Therapy - week 3 | 6.88 (0.58)
  Standard Behavior Therapy - week 4 | 6.10 (0.59)
  Modified Behavior Therapy - week 1 | 6.15 (0.63)
  Modified Behavior Therapy - week 2 | 6.38 (0.60)
  Modified Behavior Therapy - week 3 | 6.12 (0.58)
  Modified Behavior Therapy - week 4 | 6.09 (0.58)

13. Secondary Outcome: IOWA Oppositional-defiant Scale - Counselor
Description: At the end of each treatment week counselors rated each child's overall oppositional-defiant behavior during the week. Rating were completed using Likert scales that ranged from 0 ("not at all") to 3 ("very much"). Items were summed to compute a scale score with a theoretical range of 0 to 15.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
units on a scale
  Standard Behavior Therapy - week 1 | 4.55 (0.56)
  Standard Behavior Therapy - week 2 | 4.99 (0.58)
  Standard Behavior Therapy - week 3 | 4.47 (0.56)
  Standard Behavior Therapy - week 4 | 4.85 (0.58)
  Modified Behavior Therapy - week 1 | 4.20 (0.56)
  Modified Behavior Therapy - week 2 | 5.01 (0.58)
  Modified Behavior Therapy - week 3 | 4.94 (0.56)
  Modified Behavior Therapy - week 4 | 5.38 (0.58)

14. Secondary Outcome: IOWA Oppositional-defiant Scale - Parent
Description: At the end of each treatment week parents rated each child's overall oppositional-defiant behavior during the week. Rating were completed using Likert scales that ranged from 0 ("not at all") to 3 ("very much"). Items were summed to compute a scale score with a theoretical range of 0 to 15.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
units on a scale
  Standard Behavior Therapy - week 1 | 6.71 (0.70)
  Standard Behavior Therapy - week 2 | 6.99 (0.56)
  Standard Behavior Therapy - week 3 | 6.50 (0.63)
  Standard Behavior Therapy - week 4 | 6.15 (0.63)
  Modified Behavior Therapy - week 1 | 5.75 (0.75)
  Modified Behavior Therapy - week 2 | 5.80 (0.57)
  Modified Behavior Therapy - week 3 | 5.26 (0.65)
  Modified Behavior Therapy - week 4 | 5.20 (0.62)

15. Secondary Outcome: WPRF Serious Conduct Problems Scale - Counselor
Description: At the end of each treatment week counselors rated each child's serious conduct problems during the week. Rating were completed on the Weekly Problem Rating Form (Haas et al, 2011) using Likert scales that ranged from 1 ("no problem") to 7 ("serious problem"). Items were averaged to compute a scale score with a theoretical range of 1 to 7, with high scores indicating more serious problems.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
units on a scale
  Standard Behavior Therapy - week 1 | 1.71 (0.12)
  Standard Behavior Therapy - week 2 | 1.81 (0.12)
  Standard Behavior Therapy - week 3 | 1.69 (0.12)
  Standard Behavior Therapy - week 4 | 1.70 (0.12)
  Modified Behavior Therapy - week 1 | 1.66 (0.12)
  Modified Behavior Therapy - week 2 | 1.83 (0.12)
  Modified Behavior Therapy - week 3 | 1.88 (0.12)
  Modified Behavior Therapy - week 4 | 1.91 (0.12)

16. Secondary Outcome: WPRF Serious Conduct Problems Scale - Parent
Description: At the end of each treatment week parents rated each child's serious conduct problems during the week. Rating were completed on the Weekly Problem Rating Form (Haas et al, 2011) using Likert scales that ranged from 1 ("no problem") to 7 ("serious problem"). Items were averaged to compute a scale score with a theoretical range of 1 to 7, with high scores indicating more serious problems.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
units on a scale
  Standard Behavior Therapy - week 1 | 2.47 (0.19)
  Standard Behavior Therapy - week 2 | 2.48 (0.19)
  Standard Behavior Therapy - week 3 | 2.22 (0.19)
  Standard Behavior Therapy - week 4 | 1.96 (0.16)
  Modified Behavior Therapy - week 1 | 2.05 (0.21)
  Modified Behavior Therapy - week 2 | 1.94 (0.19)
  Modified Behavior Therapy - week 3 | 2.03 (0.19)
  Modified Behavior Therapy - week 4 | 2.00 (0.16)

17. Secondary Outcome: WPRF Rule Following Problems - Counselor
Description: At the end of each treatment week counselors rated each child's rule following problems during the week. Rating were completed on the Weekly Problem Rating Form (Haas et al, 2011) using Likert scales that ranged from 1 ("no problem") to 7 ("serious problem"). Items were averaged to compute a scale score with a theoretical range of 1 to 7, with high scores indicating more serious problems.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
units on a scale
  Standard Behavior Therapy - week 1 | 2.07 (0.14)
  Standard Behavior Therapy - week 2 | 2.18 (0.15)
  Standard Behavior Therapy - week 3 | 2.17 (0.15)
  Standard Behavior Therapy - week 4 | 2.19 (0.16)
  Modified Behavior Therapy - week 1 | 2.10 (0.14)
  Modified Behavior Therapy - week 2 | 2.17 (0.15)
  Modified Behavior Therapy - week 3 | 2.26 (0.15)
  Modified Behavior Therapy - week 4 | 2.30 (0.15)

18. Secondary Outcome: WPRF Rule Following Problems - Parent
Description: At the end of each treatment week parents rated each child's rule following problems during the week. Rating were completed on the Weekly Problem Rating Form (Haas et al, 2011) using Likert scales that ranged from 1 ("no problem") to 7 ("serious problem"). Items were averaged to compute a scale score with a theoretical range of 1 to 7, with high scores indicating more serious problems.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
units on a scale
  Standard Behavior Therapy - week 1 | 3.63 (0.25)
  Standard Behavior Therapy - week 2 | 3.88 (0.26)
  Standard Behavior Therapy - week 3 | 3.37 (0.25)
  Standard Behavior Therapy - week 4 | 3.47 (0.24)
  Modified Behavior Therapy - week 1 | 3.35 (0.26)
  Modified Behavior Therapy - week 2 | 3.31 (0.26)
  Modified Behavior Therapy - week 3 | 3.12 (0.26)
  Modified Behavior Therapy - week 4 | 3.31 (0.24)

19. Secondary Outcome: WPRF Overall Problems - Counselor
Description: At the end of each treatment week counselors rated each child's overall problems during the week. Rating were completed on the Weekly Problem Rating Form (Haas et al, 2011) using Likert scales that ranged from 1 ("no problem") to 7 ("serious problem"). Items were averaged to compute a scale score with a theoretical range of 1 to 7, with high scores indicating more serious problems.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
units on a scale
  Standard Behavior Therapy - week 1 | 3.42 (0.18)
  Standard Behavior Therapy - week 2 | 3.66 (0.19)
  Standard Behavior Therapy - week 3 | 3.49 (0.19)
  Standard Behavior Therapy - week 4 | 3.46 (0.18)
  Modified Behavior Therapy - week 1 | 3.36 (0.18)
  Modified Behavior Therapy - week 2 | 3.38 (0.19)
  Modified Behavior Therapy - week 3 | 3.63 (0.19)
  Modified Behavior Therapy - week 4 | 3.72 (0.18)

20. Secondary Outcome: WPRF Overall Problems - Parent
Description: At the end of each treatment week parents rated each child's overall problems during the week. Rating were completed on the Weekly Problem Rating Form (Haas et al, 2011) using Likert scales that ranged from 1 ("no problem") to 7 ("serious problem"). Items were averaged to compute a scale score with a theoretical range of 1 to 7, with high scores indicating more serious problems.
Time Frame: Weekly
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Overall Sample
Number analyzed (Participants) | 45
units on a scale
  Standard Behavior Therapy - week 1 | 3.68 (0.27)
  Standard Behavior Therapy - week 2 | 3.98 (0.26)
  Standard Behavior Therapy - week 3 | 3.57 (0.24)
  Standard Behavior Therapy - week 4 | 3.42 (0.25)
  Modified Behavior Therapy - week 1 | 3.65 (0.29)
  Modified Behavior Therapy - week 2 | 3.62 (0.26)
  Modified Behavior Therapy - week 3 | 3.43 (0.25)
  Modified Behavior Therapy - week 4 | 3.44 (0.25)

21. Secondary Outcome: How Much Did Your Child Benefit From Treatment?
Description: At the end of each treatment block parents rated their overall satisfaction with the treatment provided to their child. This item was phrased as follows: "How much did your child benefit from this treatment?". This item was rated using a Likert scale that ranged from 0 ("not at all") to 3 ("very much").
Time Frame: End of each treatment, at weeks 4 and 8
Population: Four children excluded from analyses; two excluded because of medication changes during treatment. One excluded because he was mistakenly enrolled (after collecting treatment data we learned that he did not meet all inclusion criteria). One was excluded because parent did not return completed ratings.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Overall Sample
Number analyzed (Participants) | 44
units on a scale
  Standard behavior therapy | 2.31 (0.15)
  Modified behavior therapy | 2.45 (0.15)

22. Secondary Outcome: How Much Did You (the Parent) Benefit From Treatment?
Description: At the end of each treatment block parents rated their overall satisfaction with the treatment provided to their child. This item was phrased as follows: "How much did you benefit from this treatment?". This item was rated using a Likert scale that ranged from 0 ("not at all") to 3 ("very much").
Time Frame: End of each treatment, at weeks 4 and 8
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Overall Sample
Number analyzed (Participants) | 44
units on a scale
  Standard behavior therapy | 2.36 (0.13)
  Modified behavior therapy | 2.40 (0.13)

23. Secondary Outcome: How Much Did Your Child Enjoy the Treatment?
Description: At the end of each treatment block parents rated their overall satisfaction with the treatment provided to their child. This item was phrased as follows: "How much did your child this treatment?". This item was rated using a Likert scale that ranged from 0 ("not at all") to 3 ("very much").
Time Frame: End of each treatment, at weeks 4 and 8
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Overall Sample
Number analyzed (Participants) | 44
units on a scale
  Standard behavior therapy | 1.89 (0.15)
  Modified behavior therapy | 2.12 (0.15)

24. Secondary Outcome: Would You Send Your Child to This Treatment Again?
Description: At the end of each treatment block parents rated their overall satisfaction with the treatment provided to their child. This item was phrased as follows: "Would you send your child to this treatment if you could do it over again?". This item was rated using a Likert scale that ranged from 0 ("no definitely") to 4 ("yes definitely").
Time Frame: End of each treatment, at weeks 4 and 8
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Overall Sample
Number analyzed (Participants) | 44
units on a scale
  Standard behavior therapy | 3.83 (0.06)
  Modified behavior therapy | 3.83 (0.06)

25. Secondary Outcome: Recommend Treatment?
Description: At the end of each treatment block parents rated their overall satisfaction with the treatment provided to their child. This item was phrased as follows: "Would you recommend this treatment to other parents?". This item was rated using a Likert scale that ranged from 0 ("no definitely") to 4 ("yes definitely").
Time Frame: End of each treatment, at weeks 4 and 8
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Overall Sample
Number analyzed (Participants) | 44
units on a scale
  Standard behavior therapy | 3.90 (0.04)
  Modified behavior therapy | 3.97 (0.04)

26. Secondary Outcome: Overall Satisfaction
Description: At the end of each treatment block parents rated their overall satisfaction with the treatment provided to their child. This item was phrased as follows: "Please rate your overall satisfaction with this treatment as compared with other treatment services your child has received". This item was rated using a Likert scale that ranged from 0 ("much less satisfied with this program") to 4 ("much more satisfied with this program").
Time Frame: End of each treatment, at weeks 4 and 8
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Overall Sample
Number analyzed (Participants) | 44
units on a scale
  Standard behavior therapy | 3.75 (0.07)
  Modified behavior therapy | 3.83 (0.07)

27. Secondary Outcome: Overall Effectiveness
Description: At the end of each treatment block parents rated their overall satisfaction with the treatment provided to their child. This item was phrased as follows: "Please rate how effective this treatment was in changing your child as compared with other treatment services your child has received". This item was rated using a Likert scale that ranged from 0 ("this treatment much less effective") to 4 ("this treatment much more effective").
Time Frame: End of each treatment, at weeks 4 and 8
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Overall Sample
Number analyzed (Participants) | 44
units on a scale
  Standard behavior therapy | 3.66 (0.10)
  Modified behavior therapy | 3.60 (0.10)

28. Secondary Outcome: Overall Treatment Recommendation - Counselor
Description: At end end of both treatment blocks, counselors sorted children into one of four treatment response groups: (1) responded best to standard behavior therapy; (2) responded best to modified behavior therapy; (3) responded well to both treatments; (4) did not respond to either treatment
Time Frame: End of all treatment, at week 8
Population: Four children excluded from analyses; two excluded because of medication changes during treatment. One excluded because he was mistakenly enrolled (after collecting treatment data we learned that he did not meet all inclusion criteria). One excluded because only completed one block of treatment.
Measure: Number; unit: percentage of participants
Groups:
- Overall Sample: Summer treatment program: Intensive behavioral treatment delivered in a summer camp setting. During one block of four weeks, participants received modified behavioral treatment (MBT) that emphasized rewards and de-emphasized punishments. During another block of four weeks, participants received standard behavior treatment (SBT) that balanced reward and punishment. Order of treatment blocks was counter-balanced across participants, and primary analyses were within-subject comparisons.
Arm/Group | Overall Sample
Number analyzed (Participants) | 44
percentage of participants
  Responded equally to both treatments | 34
  Responded best to standard treatment | 27
  Responded best to modified treatment | 23
  Did not respond to either treatment | 16

29. Secondary Outcome: Overall Treatment Recommendation - Parent
Description: At end end of both treatment blocks, parents selected which treatment they though was best for their child - standard behavioral treatment or modified behavioral treatment
Time Frame: End of all treatment, at week 8
Population: as for outcome 28
Measure: Number; unit: percentage of participants
Arm/Group | Overall Sample
Number analyzed (Participants) | 44
percentage of participants
  Responded best to standard treatment | 41
  Responded best to modified treatment | 59

ADVERSE EVENTS:
Description: Serious and other (Not including Serious) Adverse Events were not collected / assessed.
Arm/Group | Modified Behavior Treatment Then Standard Behavior Treatment | Standard Behavior Treatment Then Modified Behavior Treatment
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No